CLINICAL TRIAL: NCT03156231
Title: Acetazolamide for Prevention of Altitude Related Illness in Patients With Chronic Obstructive Pulmonary Disease (COPD). Randomized, Placebo-Controlled, Double-Blind Trial.
Brief Title: Effect Of Acetazolamide On Altitude Related Illness In Patients With Respiratory Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-00137
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2017-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: airway disease; bronchitis; emphysema; altitude; prevention; acetazolamide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Emphysema | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 375mg/day (capsule @125 mg: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3200m until the morning after the second night at 3200m
  Interventions: Drug: ACETAZOLAMIDE oral capsule
- PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3200m until the morning after the second night at 3200m.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ACETAZOLAMIDE oral capsule — Administration of 125mg acetazolamide in the morning, 250mg in the evening, starting 24 hours before departure to 3200m
  Arms: ACETAZOLAMIDE oral capsule
Drug: Placebo oral capsule — Administration of equally looking placebo capsules in the morning and evening, starting 24 hours before departure to 3200m
  Arms: PLACEBO oral capsule

SUMMARY:
Randomized, placebo controlled trial evaluating efficacy of acetazolamide in preventing altitude related adverse health effects (ARAHE) in lowlanders with chronic obstructive lung disease travelling from 760 m to 3200 m.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind parallel trial evaluating the efficacy of acetazolamide prophylaxis in reducing the incidence of altitude related adverse health effects (ARAHE) in lowlanders with chronic obstructive pulmonary disease travelling to altitude. Participants living in the Bishkek area, Kyrgyzstan (760m), will be transferred by car within 4h to the Tuja Ashu high altitude clinic (3200 m), and stay there for 2 days. Acetazolamide 375mg/day (or placebo), will be administered before departure at 760 m and during the stay at altitude. Outcomes will be assessed during the stay at 3200 m.

An interim analysis will be carried out when 90 patients will have completed the study or after the first year. The Peto's method will be used to correct the P-values.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age 18-75 yrs.
* COPD diagnosed according to GOLD, FEV1 40-80% predicted, SpO2 ≥92% at 750 m.
* Born, raised and currently living at low altitude (<800m).
* Written informed consent.

Exclusion Criteria:

* COPD exacerbation, very severe COPD with hypoxemia at low altitude (FEV1/FVC <0.7, FEV1 <40% predicted, oxygen saturation on room air <92% at 750 m).
* Comorbidities such as uncontrolled cardiovascular disease, i.e., unstable systemic arterial hypertension, coronary artery disease; previous stroke; OSA; pneumothorax in the last 2 months.
* Internal, neurologic, rheumatologic or psychiatric disease including current heavy smoking (>20 cigarettes per day)
* Known renal failure or allergy to acetazolamide and other sulfonamides

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Altitude related adverse health effects (ARAHE), cumulative incidence | Day 1 to 3 at 3200m
  Difference between acetazolamide and placebo group in cumulative incidence of ARAHE during the stay at 3200 m.
  ARAHE are defined as the following:
  * Moderate to severe AMS (Lake Louise score ≥3 and/or Environmental Symptoms questionnaire AMSc score ≥0.7) and/or any of the following:
  * Severe hypoxemia (SpO2 at rest <80% for >30 min or <75% for >15 min, exercise oxygen desaturation SpO2 <75% for >1 min accompanied by symptoms or signs of hypoxemia)
  * Symptomatic cardiovascular disease (arterial blood pressure systolic >200 mmHg, diastolic >110 mmHg not responding to blood pressure lowering drugs within 1 hr; chest pain with ECG signs of ischemia or new onset arrhythmia)
  * Withdrawal from the study by the decision of the independent physician for safetey reasons or by the patient

SECONDARY OUTCOMES:
Acute mountain sickness, severity | Day 1 to 3 at 3200m
  Difference between acetazolamide and placebo group in the acute mountain sickness severity assessed by the Lake Louise questionnaire.
6 min walk distance | Day 2 at 760m and 3200m
  Difference in altitude-induced change in the distance walked in 6 min between the acetazolamide and placebo group.
Perceived exertion | Day 2 at 760m and 3200m
  Difference in altitude-induced change in the perceived exertion rated with the Borg CR10 scale between the acetazolamide and placebo group
Spirometry | Day 2 at 760m and 3200m
  Difference in altitude-induced change in the spirometric variables between the acetazolamide and placebo group
Arterial blood gases | Day 2 at 760m and 3200m
  Difference in altitude-induced change in arterial oxygen partial pressure, carbon dioxide partial pressure, and pH between the acetazolamide and placebo group
Exercise endurance during constant load cycling ergometry | Day 3 at 760m and 3200m
  Difference in altitude-induced change in exercise endurance between acetazolamide and placebo group, measured by constant load cycling ergometry
Side effects | Day 1 to 3 at 3200m
  Difference between acetazolamide and placebo group in the cumulative incidence of medication side effects during the stay at 3200 m.

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schmuziger YA, Mademilov M, Buergin A, Scheiwiller PM, Mayer L, Schneider SR, Lichtblau M, Bitos K, Muralt L, Muller J, Akylbekov A, Mirzalieva G, Sooronbaev TM, Ulrich S, Bloch KE, Furian M. Nocturnal cerebral oxygenation in patients with COPD at altitude: data from a randomized clinical trial of acetazolamide. J Clin Sleep Med. 2025 Dec 1;21(12):2051-2061. doi: 10.5664/jcsm.11868. PMID 41025408
- [Derived] Christen M, Buergin A, Mademilov M, Mayer L, Schneider SR, Lichtblau M, Sooronbaev TM, Ulrich S, Bloch KE, Furian M. Electrocardiographic signs of cardiac ischemia at rest and during exercise in patients with COPD traveling to 3,100 m: data from a randomized trial of acetazolamide. Front Cardiovasc Med. 2025 Feb 6;12:1524201. doi: 10.3389/fcvm.2025.1524201. eCollection 2025. PMID 39981351
- [Derived] Furian M, Mademilov M, Buergin A, Scheiwiller PM, Mayer L, Schneider S, Emilov B, Lichtblau M, Bitos K, Muralt L, Groth A, Reiser AE, Sevik A, Sheraliev U, Marazhapov NH, Aydaralieva S, Muratbekova A, Tabyshova A, Abdraeva A, Buenzli S, Sooronbaev TM, Ulrich S, Bloch KE. Acetazolamide to Prevent Adverse Altitude Effects in COPD and Healthy Adults. NEJM Evid. 2022 Jan;1(1):EVIDoa2100006. doi: 10.1056/EVIDoa2100006. Epub 2021 Dec 22. PMID 38296630